CLINICAL TRIAL: NCT05708742
Title: The Analgesic Efficacy of Erector Spinae Plane Block in Ankle and Foot Surgery: A Randomized Controlled Study
Brief Title: Erector Spinae Plane Block and Ankle and Foot Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Hamed, Associate professor of anesthesia, Fayoum University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: D295
Record Dates: First submitted 2023-01-24; First posted 2023-02-01 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Pain; Ankle Injuries
Keywords: Erector spinae block; Ankle and foot surgery; Postoperative analgesia
MeSH Terms: conditions — Pain; Ankle Injuries | interventions — Ultrasonography; Bupivacaine; Anesthetics, Local; Saline Solution; Needles

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Apart from the anesthesiologists who performed the blocks, all patients, surgeons, and postoperative nurses remained blinded to randomization throughout the study period.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Sham Comparator): The control group underwent US-guided sham block at L4 vertebrae level with 20 ml of saline 0.9%. At the level of L4 and after skin sterilization, sham block was administered in a sitting position. Hydro dissection of the interfascial plane between the erector spinae muscle and TP was confirmed by visualizing the local anesthetic spreading in a linear pattern between the muscle and the bony acoustic shadows of the TP. Then, up to 20 ml Saline 0.9% was injected.
  Interventions: Device: Ultrasound; Drug: saline solution; Device: Needle
- ESP group (Experimental): The ESP group underwent US-guided ESP block at L4 vertebrae level with 20 ml of bupivacaine 0.25%. After skin sterilization, ESP block was administered in a sitting position. A linear US transducer was placed vertically 3 cm lateral to the midline to visualize back muscles: the trapezius above, the rhomboid major in the middle, and the erector-spinae muscle on the bottom, as well as the TPs with shimmering pleura in between. Next, 2-3 ml of 2% lidocaine was infiltrated. Hydro dissection of the interfascial plane between the erector spinae muscle and TP was confirmed by visualizing the local anesthetic spreading in a linear pattern between the muscle and the bony acoustic shadows of the TP.
  Interventions: Device: Ultrasound; Drug: Bupivacaine Hydrochloride; Device: Needle

INTERVENTIONS:
Device: Ultrasound — A linear US transducer (Phillips-Saronno Italy) was placed vertically 3 cm lateral to the midline to visualize back muscles: the trapezius above, the rhomboid major in the middle, and the erector-spinae muscle on the bottom, as well as the TPs with shimmering pleura in between.
  Other Names: Linear transducer
Drug: Bupivacaine Hydrochloride — The ESP block group underwent US-guided ESP block at L4 vertebrae level with 20 ml of bupivacaine 0.25%.
  Other Names: Local anesthetic
  Arms: ESP group
Drug: saline solution — The control group underwent the same procedure but had a sham injection (20 ml of saline).
  Other Names: Saline isotonic 0.9%
  Arms: Control group
Device: Needle — A 22-gauge short bevel needle (Spinocan, B. Braun Melsungen AG, Germany) was inserted in the cranial-caudal direction towards the TP in-plane with the US transducer until the needle touched the TP crossing all three muscles.

SUMMARY:
Regional anesthesia is commonly used in orthopedic and surgical procedures in ankle and foot surgery to manage pain. The ultrasound-guided nerve block is a safe and effective regional anesthesia technique that provides effective pain management, decreasing opioid consumption.

Postoperative pain management may be challenging and requires a multimodal approach. Regional anesthesia techniques in the pediatric ankle and foot surgery population are frequently used in postoperative pain management due to ultrasonography's increased experience and accessibility.

Erector spinae plane block (ESP) is a relatively new regional anesthesia technique that provides analgesia covering spinal nerves' dorsal and ventral rami. There are few cases reports in the literature on the use of ESP block for lower limb surgery, for which it has a promising potential for future indication.

The erector spinae plane block is a safe and effective regional anesthesia technique, which has earned new indications perioperatively since its description.

DETAILED DESCRIPTION:
This single-center study was a prospective randomized controlled trial, using parallel groups with a 1:1 allocation ratio. Eligible patients were identified by the surgeon and invited to participate in the study. If the patient wished to participate in the study, informed consent was obtained. The patient was informed of the study's nature, especially that the patient would be randomized to receive an ESPB or a sham block before the procedure. A computerized randomization program (permuted block randomization) was used to create the allocation before the beginning of the study. Research staff not involved in the recruitment process or the study's conduct randomized patients at the time of admission to the clinic. Randomization allocation was 1:1 between treatment and control groups. Apart from the anesthesiologists who performed the blocks, all patients, surgeons, and postoperative nurses remained blinded to randomization throughout the study period. The outcome parameters were recorded through a study nurse who was not involved in the patients' care.

All patients received standardized anesthesia, and all blocks were performed by 2 anesthesiologists who were trained in this technique. A large-bore intravenous (IV) line was placed, and patients received midazolam 1 to 2 mg IV for anxiolysis.

Anesthesia was induced with fentanyl 2 mcg.kg-1 and propofol 2 mg.kg-1 followed by atracurium 0.5 mg.kg-1 . After intubation, anesthesia was maintained with isoflurane (1 MAC) and atracurium 0.1mg.kg-1 as a maintenance dose every 30 min until the end of the procedure. After emerging from anesthesia, patients were transferred to the postanesthesia care unit (PACU) for a 2-h observation period. Patients were discharged from the PACU when they achieved a modified Aldrete score ≥ 9.10. Postoperative analgesia was provided in both groups immediately after surgery by PCA fentanyl pump, then oral acetaminophen 1 g four times a day. The criteria to stop the fentanyl titration protocol included satisfactory pain control, increased sedation (Ramsay sedation scale >2), decreased respiratory rate.

Statistical Analyses The sample size was estimated to achieve a power of 0.8 to detect a supposed medium effect size of 0.7 in between the two groups regarding total morphine consumption, with a 2-sided significance level of .05 and allocation ratio of 1. Thirty patients in each group were required. Allowing for a 10% loss, 34 patients were recruited in each group, for a total of 68 patients. The sample size was determined using G*Power software (version 3.1.9.7).

Descriptive statistics, including age, sex, body mass index, baseline pain scores, procedure type, traction time, and procedure time, were comparatively analyzed between the groups. Categorical data were compared with chi-squared and Fisher's exact tests as appropriate. Continuous data were compared with a 2-sided t test (for normally distributed data) and Wilcoxon rank-sum test (for non normally distributed data). For all analyses (primary and secondary measures), a P value of .05 was used to determine statistical significance. Statistical analyses were conducted using SPSS version 28 (Addinsoft, Paris, France).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 65 years, American Society of Anesthesiologists physical status classification Ι and ΙΙ; scheduled for ankle and foot surgery

Exclusion Criteria:

* Major hepatic
* severe renal impairment (creatinine > 3 or on dialysis);
* severe cardiovascular disease (ejection fraction < 35%)
* local infection at site of injection
* Any contraindication for ESP
* Known allergy to any drug used in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog score | 8 hours after operation
  0 - 10 with 0: no pain and 10: worst pain

SECONDARY OUTCOMES:
Total opioid consumption | First 24 hours postoperatively.
  in milligram
time to first analgesic request | First 24 hours postoperatively.
  from end of operation to request of analgesia due to pain
Incidence of nausea | First 24 hours postoperatively.
  yes or no
Incidence of vomiting | First 24 hours postoperatively.
  yes or no
patient satisfaction | First 24 hours postoperatively.
  1:3 with 1: very satisfied to 3: very unsatified
Incidence of local anesthetic toxicity | First 24 hours postoperatively.
  yes or no
Visual Analog score | 4 hours after operation
  0 - 10 with 0: no pain and 10: worst pain
Visual Analog score | 12 hours after operation
  0 - 10 with 0: no pain and 10: worst pain
Visual Analog score | 24 hours after operation
  0 - 10 with 0: no pain and 10: worst pain

OTHER OUTCOMES:
Age | 1 hour preoperatively
  in years
Height | 1 hour preoperatively
  in centimeter
weight | 1 hour preoperatively
  in kilogram
Sex | 1 hour postoperatively
  Female or Male

CONTACTS AND LOCATIONS:
Overall Officials: Omar S Fargahly, MD, Study Chair — Fayoum University; Rana A Abdel ghaffar, MD, Study Director — Fayoum University; Mohamed F Algyar, MD, Study Director — Kafr Elshiekh University
Locations (1):
- Fayoum University hospital, El Fayoum Qesm, Faiyum Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Diwan S, Nair A. Lumbar erector spinae plane block obtunding knee and ankle reflexes. Saudi J Anaesth. 2021 Apr-Jun;15(2):222-224. doi: 10.4103/sja.SJA_79_20. Epub 2021 Apr 1. PMID 34188648